CLINICAL TRIAL: NCT04910152
Title: A Single Arm, Open Label, Phase 1b/2 Study of Novel BET Inhibitor PLX51107 for Steroid-Refractory Acute GVHD
Brief Title: Novel BET Inhibitor PLX51107 for Steroid-Refractory Acute GVHD
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Hannah Choe, MD (Other)
Collaborators: Plexxikon (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Hannah Choe, MD, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-20273; NCI-2021-02282 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R01CA252469 (NIH)
Record Dates: First submitted 2021-04-24; First posted 2021-06-02 (Actual); Results first posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Acute Graft Versus Host Disease; Steroid Refractory Graft Versus Host Disease
MeSH Terms: interventions — PLX51107

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment for aGVHD (BRD4 inhibitor PLX51107) (Experimental): Patients receive BRD4 inhibitor PLX51107 PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: BRD4 Inhibitor PLX51107

INTERVENTIONS:
Drug: BRD4 Inhibitor PLX51107 — Given PO
  Other Names: PLX 51107; PLX-51107; PLX51107

SUMMARY:
This phase Ib/II trial studies the side effects of PLX51107 in treating steroid-refractory acute graft versus host disease (GVHD). PLX51107 is a novel, potent non-benzodiazepine structured small molecule BET inhibitor with a unique binding mode selective for BRD4 inhibition and a more tolerable side effect profile. PLX51107 may work better in treating steroid-refractory acute GVHD.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of BRD4 inhibitor PLX51107 (PLX51107) as a single agent for allogeneic transplant recipients with steroid-refractory acute graft versus host disease (GVHD).

II. To assess the pharmacokinetic (PK) and pharmacodynamic (PD) of orally administered PLX51107 in steroid-refractory acute GVHD patients.

SECONDARY OBJECTIVE:

I. To evaluate the preliminary efficacy of PLX51107 in steroid-refractory acute GVHD patients.

OUTLINE:

Patients receive BRD4 inhibitor PLX51107 orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years at the time of signing informed consent
* Steroid-refractory acute GVHD as defined as progression of acute (a)GvHD within 3-5 days of therapy onset with >= 2 mg/kg/day of prednisone equivalent OR failure to improve within 5-7 days of treatment initiation with > 1-2 mg/kg/day of prednisone equivalent OR incomplete response after more than 28 days of immunosuppressive treatment including steroids
* Recipients of ablative and reduced-intensity conditioning regimens
* Recipients of human leukocyte antigen (HLA)-matched related and unrelated, 1-allele mismatched, haploidentical, or umbilical cord blood donor grafts
* Prior lines of therapy for treatment of steroid-refractory acute GVHD are allowed. However, exposure to investigational therapies for the treatment of GVHD must be > 14 days or 5 half-lives (whichever is shorter) of first administration of study drug. For patients treated with ruxolitinib for the treatment of acute GVHD, ruxolitinib must be discontinued by at least one day prior to initiation of PLX51107
* Eastern Cooperative Oncology Group (ECOG) performance status =< 3
* Absolute neutrophil count >= 1.0 x 10^9/L for 3 consecutive days). Use of growth factor support is allowed
* Platelet count >= 50 x 10^9/L without transfusion support for 2 consecutive days
* Women of child-bearing potential must have a negative serum pregnancy test at Screening and must agree to use an effective form of contraception from the time of the negative pregnancy test up to 6 months after the last dose of study drug. Effective forms of contraception include abstinence, hormonal contraceptive in conjunction with a barrier method, or a double barrier method. Women of non-child-bearing potential may be included if they are either surgically sterile or have been postmenopausal for >= 1 year
* Fertile men must agree to use an effective method of birth control during the study and for up to 6 months after the last dose of study drug

Exclusion Criteria:

* Prior exposure to a bromodomain inhibitor
* Evidence of chronic GVHD
* Evidence of active relapse of disease
* Exposure to other investigational or anti-cancer therapies (not for GVHD) within 28 days or 5 half-lives (whichever is shorter) of first administration of study drug
* Active, uncontrolled bacterial, fungal, or viral infection
* Known or suspected allergy to the study drug
* Clinically significant cardiac disease, defined as:

  * Clinically significant cardiac arrhythmias, including bradyarrhythmia, and/or a need for anti-arrhythmic therapy (excluding beta blockers or digoxin). Individuals with controlled atrial fibrillation are not excluded
  * Fridericia-corrected QT interval (QTcF) >= 450 ms (male) or >= 470 ms (female) at screening
  * History of clinically significant cardiac disease or congestive heart failure greater than New York Heart Association Class II. Subjects must not have unstable angina (angina symptoms at rest) or experienced either new-onset angina within the last 3 months or myocardial infarction (MI) within the last 6 months unless it was due to the underlying disease and there has been appropriate revascularization. Individuals with ambiguous troponin levels that are not diagnostic of an MI should be discussed with the principal investigator (PI) prior to enrollment
  * Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis, or pulmonary embolism within the 6 months before start of study medication (except for catheter-related venous thrombosis
* Inability to take oral medication or significant nausea and vomiting, malabsorption, or significant small bowel resection that, in the opinion of the Investigator, would preclude adequate absorption
* Active thrombotic microangiopathy (TMA)
* Women who are either pregnant or breast feeding
* Measured or calculated (Cockcroft-Gault formula) creatinine clearance (CrCl) < 45 mL/min
* Prothrombin time or international normalized ratio > 1.5 x upper limit of normal (ULN)
* Activated partial thromboplastin time > 1.5 x ULN
* Requiring mechanical ventilation or vasopressor support
* Subject is participating in any other therapeutic clinical study (observational or registry studies are allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Choe, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment for aGVHD (BRD4 Inhibitor PLX51107)
Started (Enrolled) | 2
Received Treatment | 1
Completed | 1
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment for aGVHD (BRD4 Inhibitor PLX51107)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Time Frame: Up to 28 days
Population: Maximum tolerated dose was not able to be determined due to low accrual number.
Arm/Group | Treatment for aGVHD (BRD4 Inhibitor PLX51107)
Number analyzed (Participants) | 0

2. Primary Outcome: Incidence of Adverse Events Grade 3 and 4
Description: Adverse events by grade will be summarized. The occurrence of grade 3+ adverse events according to Common Terminology Criteria for Adverse Events will be summarized as well. Adverse events will initially be reviewed regardless of attribution, but also according to whether adverse events are possibly, probably, or definitely related to treatment.
Time Frame: Up to 6 months
Measure: Number; unit: participants
Arm/Group | Treatment for aGVHD (BRD4 Inhibitor PLX51107)
Number analyzed (Participants) | 1
participants
  Grade 1 Adverse Events : Bloating | 1
  Grade 1 Adverse Events : Confusion | 1
  Grade 1 Adverse Events : Dyspnea | 1
  Grade 2 Adverse Events : Creatinine Increased | 1
  Grade 2 Adverse Events : Neutrophil Count Decreased | 1
  Grade 3 Adverse Events : Anemia | 1
  Grade 3 Adverse Events : Creatinine Increased | 1
  Grade 3 Adverse Events : Neutrophil Count Decreased | 1
  Grade 3 Adverse Events : Adult Respiratory Distress Syndromre | 1
  Grade 3 Adverse Events : Upper Gastrointestinal Hemorrhage | 1
  Grade 3 Adverse Events : White Blood Cell Decreased | 1
  Grade 4 Adverse Events : Platelet Count Decreased | 1
  Grade 4 Adverse Events : White Blood Cell Decreased | 1

3. Secondary Outcome: Complete Response (CR)
Description: The proportion of CR with a 95% confidence interval will be reported, assuming a binomial distribution.
Time Frame: At day 28
Population: Complete response data was not collected due to low accrual numbers
Arm/Group | Treatment for aGVHD (BRD4 Inhibitor PLX51107)
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Response Rate
Description: The overall response rate (ORR) will include CR and partial response (PR), while mixed response (MR) and no response (NR) will be classified as no response. The ORR will be similarly analyzed as CR.
Time Frame: At day 28
Population: Overall response data was not collected due to low accrual numbers.
Arm/Group | Treatment for aGVHD (BRD4 Inhibitor PLX51107)
Number analyzed (Participants) | 0

5. Secondary Outcome: Non-relapse Mortality (NRM)
Description: The cumulative incidence curve accounting for competing risks will be generated to estimate the cumulative incidence of NRM rate at 6 months. The comparison in NRM between patient subgroups may be explored graphically.
Time Frame: From the date of starting PLX51107 to date of death with the competing risk as death due to disease, assessed at 6 months
Population: NRM data was not collected due to low accrual numbers
Arm/Group | Treatment for aGVHD (BRD4 Inhibitor PLX51107)
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Pharmacokinetics (PK) Analysis
Description: Pharmacokinetics (PK) for target exposure of AUC0-24 8300 ng•hr/mL
Time Frame: Up to 6 months
Population: PK analysis data was not collected due to low accrual numbers
Arm/Group | Treatment for aGVHD (BRD4 Inhibitor PLX51107)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Patients were evaluated for adverse events using the NCI CTCAE version 5.0 from the start of study up to 1 year, 5 months.
Arm/Group | Treatment for aGVHD (BRD4 Inhibitor PLX51107)
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment for aGVHD (BRD4 Inhibitor PLX51107) (N=1)
Multi-organ failure (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment for aGVHD (BRD4 Inhibitor PLX51107) (N=1)
Bloating (Gastrointestinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Creatinine Increased (Investigations) | 1 (1)
White Blood Cell Decreased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Platelet Count Decreased (Investigations) | 1 (1)
Neutrophil Count Decreased (Investigations) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-17): https://cdn.clinicaltrials.gov/large-docs/52/NCT04910152/Prot_SAP_001.pdf
  • Informed Consent Form (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/52/NCT04910152/ICF_000.pdf